CLINICAL TRIAL: NCT07406386
Title: Integrating Halotherapy Into Preseason Training Improves Respiratory and Aerobic Performance in Elite Female Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, Director, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/2-3
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Aerobic Performance; Respiratory Function; Athletic Performance; Respiratory Muscle Strength; Elite Female Athletes; Halotherapy
Keywords: Halotherapy; Elite female soccer players; Respiratory muscle strength; Pulmonary function; Aerobic capacity; Non-pharmacological intervention
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Halotherapy sessions were conducted in a controlled halochamber using a dry salt aerosol generator. Sessions lasted 45 minutes and were performed three times per week for 12 weeks. Aerosol concentration was maintained at approximately 20 mg/m³ with particle size <5 microns. Environmental conditions were controlled (temperature 20-24°C, humidity 40-60%).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Halotherapy Group (Experimental): Participants followed the standard preseason soccer training program and additionally received halotherapy. Halotherapy sessions were conducted in a controlled halochamber using a dry salt aerosol generator. Sessions lasted 45 minutes and were performed three times per week for 12 weeks. Aerosol concentration was maintained at approximately 20 mg/m³ with particle size <5 microns. Environmental conditions were controlled (temperature 20-24°C, humidity 40-60%).
  Interventions: Other: Halotherapy Group; Other: Control
- CONTROL (No Intervention): Participants followed the same standard preseason soccer training program without halotherapy.

INTERVENTIONS:
Other: Halotherapy Group — Participants followed the standard preseason soccer training program and additionally received halotherapy.
  Halotherapy sessions were conducted in a controlled halochamber using a dry salt aerosol generator. Sessions lasted 45 minutes and were performed three times per week for 12 weeks. Aerosol concentration was maintained at approximately 20 mg/m³ with particle size <5 microns. Environmental conditions were controlled (temperature 20-24°C, humidity 40-60%).
  Arms: Halotherapy Group
Other: Control — Participants followed the same standard preseason soccer training program without halotherapy.
  Arms: Halotherapy Group

SUMMARY:
This randomized controlled trial aimed to investigate the effects of a 12-week halotherapy intervention on respiratory muscle strength, pulmonary function, aerobic capacity, and intermittent running performance in elite female soccer players. Participants were randomly assigned to either a halotherapy group or a control group. Both groups followed the same preseason soccer training program, while the halotherapy group additionally received regular halotherapy sessions. Pre- and post-intervention assessments included spirometric measurements, respiratory muscle strength, estimated VO₂max, and Yo-Yo Intermittent Recovery Test Level 1 performance.

DETAILED DESCRIPTION:
Aerobic capacity and respiratory efficiency are critical determinants of performance in elite soccer. Halotherapy, a non-pharmacological intervention involving inhalation of dry salt aerosol in a controlled environment, has been shown to improve pulmonary health in clinical populations; however, evidence in athletic populations remains limited.

This randomized parallel-group trial was conducted during the preseason period of the Turkish Women's First League. Twenty-eight elite female soccer players were randomly allocated to a halotherapy group or a control group. Both groups completed an identical 12-week soccer training program. In addition to training, the halotherapy group underwent 45-minute halotherapy sessions three times per week in a controlled halochamber environment.

Outcome measures included maximal inspiratory and expiratory pressures (MIP, MEP), pulmonary function parameters (FVC, FEV₁, PEF, MVV), aerobic capacity estimated via the Yo-Yo Intermittent Recovery Test Level 1, and total distance covered in the Yo-Yo test. Measurements were collected before and after the intervention period. The study aimed to determine whether halotherapy provides additive benefits to standard soccer training in elite female athletes.

ELIGIBILITY:
Inclusion Criteria:

* Female soccer players aged 18-30 years
* Competing in the Turkish Women's First League
* Minimum of 5 years of competitive soccer experience
* Regular training ≥10 hours per week
* Free from injury at study entry
* Non-smokers
* Not using chronic medication
* Provided written informed consent

Exclusion Criteria:

* Presence of respiratory, cardiovascular, or metabolic disease
* Current musculoskeletal injury
* Smoking
* Pregnancy
* Use of medications affecting respiratory or cardiovascular function

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female soccer players aged 18-30 years Competing in the Turkish Women's First League Minimum of 5 years of competitive soccer experience
Enrollment: 28 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Maximal Expiratory Pressure (MEP) | 12 week
  Expiratory muscle strength measured using a portable respiratory pressure meter.
Maximal Inspiratory Pressure (MIP) | 12 week
  Inspiratory muscle strength measured using a portable respiratory pressure meter.
Aerobic Capacity (VO₂max estimate) | 12 week
  VO₂max estimated using the Yo-Yo Intermittent Recovery Test Level 1.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | 12 week
  Measured by spirometry.
Forced Expiratory Volume in 1 Second (FEV₁) | 12 weeks
  Measured by spirometry.
Peak Expiratory Flow (PEF) | 12 week
  Measured by spirometry.
Yo-Yo Intermittent Recovery Test Level 1 Distance | 12 week
  VO₂max estimated using the Yo-Yo Intermittent Recovery Test Level 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Gümüşhane, Trabzon, Ordu, Giresun, Rize, Artvin, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves a small sample of elite athletes from a single professional team, which may increase the risk of indirect participant identification. Additionally, the informed consent obtained from participants did not include explicit permission for public sharing of individual-level data. Data are therefore available only in aggregated form to protect participant confidentiality.